CLINICAL TRIAL: NCT07402447
Title: Effect of Combined Quadriceps and Calf Strengthening Program on Gait, Functionality, and Sleep Quality in Knee Osteoarthritis Patients
Brief Title: Effect of Combined Quadriceps and Calf Strengthening Program on Gait in Knee Osteoarthritis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RiphahIU - Sarah Rehman
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
Keywords: Calf Strengthening; Gait; Sleep quality; Quadriceps Strengthening
MeSH Terms: conditions — Osteoarthritis, Knee; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Combined Quadriceps and Calf Strengthening) (Experimental): The experimental group will receive physiotherapy treatment consisting of the application of a heating pad for 10 minutes, followed by Grade II joint mobilization, quadriceps strengthening exercises, and calf strengthening exercises
  Interventions: Other: Group A (Combined Quadriceps and Calf Strengthening)
- Group B (Conventional) (Active Comparator): The control group will receive conventional physiotherapy treatment, which included the application of a heating pad for 10 minutes, followed by Grade II joint mobilization, and quadriceps strengthening exercises.
  Interventions: Other: Group B( Conventional)

INTERVENTIONS:
Other: Group A (Combined Quadriceps and Calf Strengthening) — During weeks 1-2, Group A will receive a heating pad for 10 minutes followed by Grade II joint mobilization. This will be followed by strengthening exercises including quadriceps strengthening in the form of straight leg raises, quadriceps sets, and leg extension exercises with 1 kg weight. Calf strengthening exercises will also be performed, including standing heel raises, seated calf raises, and standing single heel raises with support. All exercises will be initially performed with 10 repetitions and 1 set.
  During weeks 3-4, the exercise protocol will progress by increasing the repetitions to 12, sets to 2, and external resistance to 1.5 kg.
  During weeks 5-6, further progression will be made by increasing the repetitions to 15, sets to 3, and external resistance to 2 kg.
  Arms: Group A (Combined Quadriceps and Calf Strengthening)
Other: Group B( Conventional) — During weeks 1-2, Group B will receive a heating pad for 10 minutes followed by Grade II joint mobilization. This will be followed by quadriceps strengthening in the form of straight leg raises, quadriceps sets, and leg extension exercises with 1 kg weight. All exercises will be initially performed with 10 repetitions and 1 set.
  During weeks 3-4, the exercise protocol will progress by increasing the repetitions to 12, sets to 2, and external resistance to 1.5 kg.
  During weeks 5-6, further progression will be made by increasing the repetitions to 15, sets to 3, and external resistance to 2 kg.
  Arms: Group B (Conventional)

SUMMARY:
The aim of this study is to determine the effects of a combined quadriceps and calf strengthening program on gait, strength, pain, disability, functional mobility, and sleep quality in patients with knee osteoarthritis. A randomized controlled trial will be conducted at Hayatabad Medical Complex, Peshawar. A total of 52 participants aged 40-60 years with grade 2-3 knee osteoarthritis will be recruited using non-probability convenience sampling and randomly allocated into experimental and control groups. Outcome measures include Kinovea software for gait analysis, hand-held dynamometer for strength, Numeric Rating Scale for pain, WOMAC for disability, Timed Up and Go test for function, and Pittsburgh Sleep Quality Index for sleep quality. Data will be analyzed using SPSS version 27 employing repeated measures ANOVA and mixed-way ANOVA.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a chronic, progressive degenerative condition commonly affecting older adults and is a major cause of disability. It is characterized by degeneration of articular cartilage, subchondral bone changes, and synovial inflammation. KOA results in pain, stiffness, impaired balance, reduced physical function, and diminished quality of life, leading to significant psychological and socioeconomic burden. Knee osteoarthritis (KOA) develops due to several factors including mechanical stress, obesity, joint injury, aging-related cartilage wear and tear, genetic predisposition, and low-grade inflammation that damages the cartilage.

Physical therapy is a key component of KOA management and focuses on pain reduction, restoration of joint mobility, and improvement in functional ability and quality of life through exercises such as quadriceps strengthening, gait and balance training, and aerobic or aquatic exercises. Quadriceps strengthening helps stabilize the knee joint, reduce abnormal loading, and improve shock absorption, thereby decreasing joint stress during daily activities.

In addition to quadriceps weakness, patients with KOA commonly exhibit reduced calf muscle strength compared to healthy individuals. The calf muscles, particularly the gastrocnemius, play an important role in knee stabilization, load absorption, and functional movements such as walking. Altered gastrocnemius activation during weight-bearing activities can negatively affect knee biomechanics and contribute to disease progression. Muscle strengthening exercises have been shown to improve muscle strength, balance, and reduce joint inflammation in KOA patients.

Literature review: In a study carried out by Paul DeVita et al in 2018 weaker quadriceps increased the risk and progression of KOA, while strengthening the quadriceps improves pain, physical function, and quality of life by providing better knee stability and reducing joint stress.

A 2020 study by Ali M. Alshami et al. reported that compared to healthy adults, calf muscle weakness and atrophy is common in patients with KOA, with muscle strength notably decreased despite flexibility and girth not being significantly affected to be.

Zhanliang Tan et al in 2025 stated that HKE targeting gastronomies muscle effectively and safely alleviated knee pain and restored function.

A systemic review by Disha D hedge et al in 2025 states that Quadriceps strengthening as a part of lower extremity strengthening is effective in reducing pain in KOA. Emine Kiyak (2018) reported that about 81% of KOA patients significant difficulties in maintaining sleep. Patients with KOA suffered from night pain, which significantly disrupted sleep and contributed to poorer overall sleep quality, ultimately diminishing quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female
* Participants aged 40-60years.
* Diagnosed with grade 2 and 3 of knee osteoarthritis according to Kellgren-Lawrence
* Quads manual muscle grading <4
* Ability to understand and comply with exercise instructions.

Exclusion Criteria:

* History of recent knee surgery or trauma in the past six months.
* Inflammatory joint diseases (e.g., rheumatoid arthritis, gout).
* Severe cardiovascular or neurological disorders.
* Uncontrolled hypertension or diabetes.
* Participation in other physiotherapy or pharmacological interventions for knee OA during the study period.
* Cognitive impairment or inability to follow commands

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Temporo-spatial Gait | from baseline to 6 weeks
  Gait parameters will be measured by Kinovea Software.A video of the gait will be recorded and then evaluated with kinovea.
Quadriceps Strength | from baseline to 6 weeks
  the Hand Held Dynamometer will be used to asses the strength of quadriceps
Calf Strength | from baseline to 6 weeks
  the Hand Held Dynamometer will be used to asses the strength of Calf

SECONDARY OUTCOMES:
Knee Pain | from baseline to 6 weeks
  Pain will be assessed using Numeric Rating Scale(NRS). it is an 11-point scale comprising a number from 0 through 10; 0 indicates "no pain", and 10 indicates the "worst imaginable pain".
knee Disability | from baseline to 6 weeks
  it will be assessed using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), . It consists of 24 items in subscale measuring pain, stiffness and physical function.
knee Function | from baseline to 6 weeks
  Time up and Go test will be used, TUG is an easy and quick test to assess the patient's functional mobility
Sleep Quality | from baseline to 6 weeks
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality. the PSQI measures seven domains of sleep quality: subjective sleep quality, sleep latency (time to fall asleep initially), sleep duration, sleep efficiency (percent of time in bed spent asleep), sleep disturbances, use of sleep medications, and daytime dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, PHD, Principal Investigator — Riphah International University
Locations (1):
- Hayatabad Medical Complex, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No